CLINICAL TRIAL: NCT03954821
Title: Effect of the Prefabricated Plantar Insoles to Control Pronation Measured With Foot Posture Index
Brief Title: How Prefabricated Plantar Insoles Can Reduce the Pronation
Status: Completed | Type: Observational
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, María Victoria Cáceres, Associated teacher of University of Extremadura, University of Extremadura
Other Study IDs: UExtremadura
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Flat Feet
Keywords: Foot posture index, foot pronation ,foot orthoses
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: control group in which all of them present pronated foot without tratment
- experimental group: Group in which they have been treated with prefabricated plantar insoles to stop pronation
  Interventions: Device: prefabricated insoles

INTERVENTIONS:
Device: prefabricated insoles
  Groups: experimental group

SUMMARY:
Pronation is a very common foot deformity in population. Plantar insoles are one way to treat it, and even correct it, but there are several kind of treatments. In this study we try to prove if prefabricated foot insoles are a solution to correct pronation in adults. It has been tested by Foot Posture Index, that it is an objetive clinical test to measure the posture of feet. Foot is clasified in supinated , pronated and neutral.

DETAILED DESCRIPTION:
Nowadays several treatments have been described to treat pronation foot posture, althought these ones heven´t proved objetively the improvement and progression of foot deformity like "Foot Posture Index" does,. Foot pronation during walking is a physiological movement at the beginning of stance phase. It is a needed mechanism which allows the lower limb muscles to support the reaction forces from the ground and to give the forefoot wider range of movement . When there is pronation movement in weight bearing of subtalar joint, the calcaneus does a movement of eversión while talus does a plantarflexion and movement of aduction .The movement is raised due to the paralelism of midfoot joints and the forefoot is forced to compensate the rearfoot position, gettting into dorsiflexion and abduction which leads to a flattening of the medial arch. it is known pronation or flatfoot. Pronation movement is a pathology when it happens during the second part of the stance phase, the 25% at the beginning or when deformity is abnormal provoking an excessive rearfoot eversion with flattenig of the medial arch which will lead to a lower limb misalignment . This doesn´t allow the foot to be a rigid part needed to propulsion phase, so muscles must work excessively to give balance. The pronated foot etiology can be congenital or laxity or due to triceps sural shortening, or functional etiology like varus forefoot, metatarsus aductus or tibial posterior insufficiency. There are some secundary painful pathologies which are the most frequent reason of podiatric appointment.. Plantar fascitis is one of the pathologies, and adquired deformities like Hallux Abductus Valgus, Hallux Límitus/Rigidus and other lower limb deformities like medial compatiment ostheoartritis of knee or patellofemoral syndrome.

Pronated foot can be defined like a foot that has rearfoot eversion and medial protusion of the head of talus, forefoot abduction, flatted medial arch and joint movement greater. This shows a flat foot aspect, depending on the grades of pronation deformity that pacient presents. Both situations are linked and their behaviour are functionally similar.

Attending on consequences and the pathologies derivated of this deformity there are some treatments to stop it and avoid structural alterations of leg and foot. For instance, hallux abductus Valgus, the pathological pronation is the first ray´s extrinsic ethilogic factor, both frequency and capacity to produce pathology.

The compensation of pathological pronation of rearfoot is important to control the deformity evolution. Is commonly accepted by podiatric scientific community that control of pronation can avoid the deformity progression when it is presented (or this progression was slower) and avoid when it wasn´t present yet. Foot Posture Index is a clinical diagnostics tool compounds by 6 criteria that allow to asses reliability the weightbearing foot posture. It is a inexpensive and simple method that doesn´t imply risks to people.

ELIGIBILITY:
Inclusion Criteria:

* feet without symptom
* not present joint deformities to difficult the right measure of them
* aged between 18 to 50 years

Exclusion Criteria:

* don´t have degenerative ostheoarticular deformities
* don´t have surgery iinterventions of lower limbs
* balance problems
* painful keratopaties or plantar warts that difficults stance phase
* use of others orthopaedics treatements (plantar insoles)
* don´t be able to step correctly and coordinated on platform to inspect the foot posture

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 'Participant were pupils of Podiatric, Nursing, Forestry and Economic grades of University of Extremadura in Plasencia Campus, Spain. All of the came to Podiatric University Clinic Of University of Extremadura, Spain to be recruided in the present study. After to be informed of the features and targets of this study, they were be given an informed consent, answering the doubts. All of them signed the informed consent and they were asked to be engaged to use the right shoes with plantar insoles all the week , 8 hours at least for 6 months.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Foot Posture Index | 5 minutes total assessment
  Foot Posture Index is a diagnostic tool to measure the foot posture while it is weightbearing. The Foot Posture Index is a 6-item foot posture assessment with the subject standing relaxed in a bipedal position, The 6 items of FPI include talar head palpation, curves above and below the lateral melleoli, calcaneal angle, talonavicular bulge, medial longitudinal arch and forefoot to rearfoot alignment. Each item was scored on a 5-point scale between -2 and +2 and provides a total sum of all items between -12 (highly supinated) and +12(highly pronated).

CONTACTS AND LOCATIONS:
Overall Officials: Julian F Garcia, Nursing, Study Director — University of Extremadura

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barton CJ, Levinger P, Crossley KM, Webster KE, Menz HB. Relationships between the Foot Posture Index and foot kinematics during gait in individuals with and without patellofemoral pain syndrome. J Foot Ankle Res. 2011 Mar 14;4:10. doi: 10.1186/1757-1146-4-10. PMID 21401957
- [Background] Benhamú S (2011). Factores pododólogicos predictivos de la laxitud ligamentosa en la población adulta [Tesis doctoral]. Departamento de Podología. Sevilla, Universidad de Sevilla.
- [Background] Cornwall MW, McPoil TG. Relationship between static foot posture and foot mobility. J Foot Ankle Res. 2011 Jan 18;4:4. doi: 10.1186/1757-1146-4-4. PMID 21244705
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Edwards MR, Jack J, Singh SK (2008). Tibialis posterior dysfunction. CurrOrthop 22(3):185-192.
- [Background] Fuller EA. The windlass mechanism of the foot. A mechanical model to explain pathology. J Am Podiatr Med Assoc. 2000 Jan;90(1):35-46. doi: 10.7547/87507315-90-1-35. PMID 10659531
- [Background] Irving DB, Cook JL, Young MA, Menz HB. Obesity and pronated foot type may increase the risk of chronic plantar heel pain: a matched case-control study. BMC Musculoskelet Disord. 2007 May 17;8:41. doi: 10.1186/1471-2474-8-41. PMID 17506905
- [Background] Levinger P, Murley GS, Barton CJ, Cotchett MP, McSweeney SR, Menz HB. A comparison of foot kinematics in people with normal- and flat-arched feet using the Oxford Foot Model. Gait Posture. 2010 Oct;32(4):519-23. doi: 10.1016/j.gaitpost.2010.07.013. Epub 2010 Aug 8. PMID 20696579
- [Background] Michaud T (1996). Foot orthoses and other forms of conservative foot cares. Massachusetts: Williams and Wilkins.
- [Background] Nielsen RG, Rathleff MS, Moelgaard CM, Simonsen O, Kaalund S, Olesen CG, Christensen FB, Kersting UG. Video based analysis of dynamic midfoot function and its relationship with Foot Posture Index scores. Gait Posture. 2010 Jan;31(1):126-30. doi: 10.1016/j.gaitpost.2009.09.012. Epub 2009 Oct 24. PMID 19854653
- [Background] Razeghi M, Batt ME. Foot type classification: a critical review of current methods. Gait Posture. 2002 Jun;15(3):282-91. doi: 10.1016/s0966-6362(01)00151-5. PMID 11983503
- [Background] Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: the Foot Posture Index. Clin Biomech (Bristol). 2006 Jan;21(1):89-98. doi: 10.1016/j.clinbiomech.2005.08.002. Epub 2005 Sep 21. PMID 16182419
- [Background] Reina M, Lafuente G, Munuera PV. Efecto de las Ortesis Plantares en las Mujeres con Hallux Abductus Valgus Leve y Moderado en Estática. Rev Esp Podol 2010; 21(5): 170-175.
- [Background] Rodríguez E. Estudio de los Efectos de los Soportes Plantares en la prevención y/o tratamiento del HAV. Rev Esp Podol 1993; 4(7): 323-330.
- [Background] Sánchez Rodríguez R (2011). Influencia del índice de Postura del pie en las presiones plantares durante la marcha. [Tesis doctoral]. Departamento de Enfermería. Plasencia, Universidad de Extremadura.
- [Background] Sánchez Rodríguez R, Martínez Nova A, Escamilla Martinez E, Gómez Martín B (2010). Patrones de presión plantar según el Índice de Postura del Pie. El peu 30(4):184-192.
- [Background] Sammarco VJ, Nichols R. Orthotic management for disorders of the hallux. Foot Ankle Clin. 2005 Mar;10(1):191-209. doi: 10.1016/j.fcl.2004.09.003. PMID 15831266
- [Background] Scott G, Menz HB, Newcombe L. Age-related differences in foot structure and function. Gait Posture. 2007 Jun;26(1):68-75. doi: 10.1016/j.gaitpost.2006.07.009. Epub 2006 Sep 1. PMID 16945538
- [Background] Teyhen DS, Stoltenberg BE, Collinsworth KM, Giesel CL, Williams DG, Kardouni CH, Molloy JM, Goffar SL, Christie DS, McPoil T. Dynamic plantar pressure parameters associated with static arch height index during gait. Clin Biomech (Bristol). 2009 May;24(4):391-6. doi: 10.1016/j.clinbiomech.2009.01.006. Epub 2009 Feb 25. PMID 19246138